CLINICAL TRIAL: NCT00975351
Title: Estimation of Plasma Folate Apparent Volume of Distribution in Adults
Acronym: FOLCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IFR4/2008; 08/H0310/154
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: folates; 5-methyltetrahydrofolic acid; pharmacokinetics; bioavailability; biotransformation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV dose of 5-methyltetrahydrofolic acid (Experimental): IV test dose of 13C5-labelled 5-methyltetrahydrofolic acid to all eligible volunteers, followed by regular blood samplings over 2hr period taken via a cannula.
  Interventions: Dietary Supplement: 13C5-labelled 5-methyltetrahydrofolic acid

INTERVENTIONS:
Dietary Supplement: 13C5-labelled 5-methyltetrahydrofolic acid — one intravenous bolus dose of no more than 500nmole 13C5-labelled 5-methyltetrahydrofolic acid, followed by multiple blood samplings at regular time intervals. Total 2hr "intervention".
  Other Names: 13C5-labelled 5 methyltetrahydrofolic acid, calcium salt; 6S-5-CH3-H4-Pte[13C5] Glu-Ca

SUMMARY:
The aim of this study is to calculate the plasma apparent volume of distribution of natural folate to give a more accurate value for use in a mathematical model of apparent folate absorption.

DETAILED DESCRIPTION:
Bioavailability is a major determinant of nutritional status. In order to determine a safe level of folate fortification, its bioavailability must be assessed, so that risk-benefit analysis can be carried out. Recently, a mathematical model of folate true absorption which takes into account the liver first pass was devised (ref 1). In this model, the volume of distribution is a convenient method for describing how well a nutrient is removed from plasma and distributed into tissues.

In this study, volume of distribution will be more accurately estimated using an intravenous dose of labelled (13C5) dose of natural folate (5-methyltetrahydrofolic acid) in healthy adults aged 18-65, over a wide body mass index (BMI) range.

Healthy adults will be given an IV dose of a small amount of 13C5 5-methyltetrahydrofolic acid, and blood samples will be taken at regular time points via a cannula over a 2hr time period.

The primary objective is to estimate the sampled plasma pool volume of distribution in order to quantify the fraction of any folate test dose, or folate metabolites, appearing in systemic plasma circulation in future studies of bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged 18-65
* Body mass index above 19.5 and below 40
* Smokers and non-smokers
* Participation in the FolGene study

Exclusion Criteria:

* Pregnancy or been pregnant in last 12 months
* History of fits, seizures or blackouts
* Parallel participation in other research projects which invole dietary intervention and/or sampling of biological fluids/material which study nurses advice would affect either wellbeing of volunteer or the study data, apart from participation in the FolGene study
* Any person related to or living with a member of the study team
* Participation in another research project which involves blood sampling within the last 4 months unless total amount blood combined from both studies is less than 470ml
* Had donated blood within 16 weeks of starting the study
* Prescribed medication for epilepsy/seizures
* Diabetics
* History of any gastrointestinal disorder requiring medical treatment
* Any long term medical condition requiring active treatment which may affect volunteers wellbeing or the study data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Estimation of sampled plasma pool volume of distribution for natural folates | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Finglas, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Background] Wright AJ, Finglas PM, Dainty JR, Wolfe CA, Hart DJ, Wright DM, Gregory JF. Differential kinetic behavior and distribution for pteroylglutamic acid and reduced folates: a revised hypothesis of the primary site of PteGlu metabolism in humans. J Nutr. 2005 Mar;135(3):619-23. doi: 10.1093/jn/135.3.619. PMID 15735104